CLINICAL TRIAL: NCT00230555
Title: The MOM Program at the Children's Hospital of Philadelphia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2001-4-2388
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2005-10-03 (Estimated); Status verified 2005-04

CONDITIONS: Child Development
Keywords: child, preschool; environment; intelligence

INTERVENTIONS:
Behavioral: professional support model

SUMMARY:
The purpose of the MOM Program is to promote child development by helping families become more competent in accessing and using available resources. The program focuses are childhood immunizations, Early Intervention services, lead screening, Early Head Start and Head Start enrollment. The hypothsis is that children receiving the intervention will participate in more of the public services and primary healthcare activities which have been shown to be effective in improving their development.

DETAILED DESCRIPTION:
The MOM Program is a 3 year randomized controlled trial of mothers and newborns. At enrollment subjects are given a questionnaire to assess self efficacy and a non-verbal test of intelligence. Program personnel are blind to the results of this testing. Test results will be used in data analysis at the end of the study to compare outcomes of the intervention and control groups and to assess how mothers with impaired cognitive ability have benefited from participation in the study.The Intervention consists of frequent phone calls and home visits to encourage mothers to have their babies immunized on schedule and to participate in needed developmental and educational services. At 33 months of age all children receive a developmental assessment.

ELIGIBILITY:
Inclusion Criteria: mothers from West and South Philadelphia who have given birth on the post-partum unit at the Hospital of the University of Pennsylvania during the six month enrollment period from July, 2001 to Jan, 2002..

-

Exclusion Criteria: women or infants who are critically ill, those involving multiple births (ie twins), and women who are solely non-English speaking.

-

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300
Dates: Start 2001-07; Study Completion 2004-11

PRIMARY OUTCOMES:
child intelligence, 33 months of age

SECONDARY OUTCOMES:
At child age 33 months: maternal intelligence
At child age 33 months:caregiver depression
At child age 33 months: childhood immunization completion At child age 33 months: Early Intervention usage

CONTACTS AND LOCATIONS:
Overall Officials: Donald F Schwarz, M.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States